CLINICAL TRIAL: NCT07006233
Title: A Novel Dietary Approach to Manage Symptoms of Narcolepsy and Idiopathic Hypersomnia
Brief Title: A Novel Approach to Manage Symptoms of Narcolepsy and Idiopathic Hypersomnia
Acronym: COMPANION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Woolcock Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPANION; 316-SR-23 (Other Grant/Funding Number: American Academy of Sleep Medicine Foundation)
Record Dates: First submitted 2025-05-05; First posted 2025-06-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Hypersomnia; Narcolepsy Type 1 (NT 1); Narcolepsy Type 2 (NT2)
Keywords: keto diet; ketogenic; keto; whole food diet; narcolepsy; idiopathic hypersomnia; low carb; hypersomnolence; diet; dietary intervention; diet intervention
MeSH Terms: conditions — Idiopathic Hypersomnia; Narcolepsy; Disorders of Excessive Somnolence | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: A prospective mixed methods clinician led randomised controlled hybrid type 1 study
Who Masked: Outcomes Assessor
Masking Description: Blinding: Single-blinded study (assessor for baseline and post-intervention data blinded).
  Interviewers for semi-structured interviews will also be blinded (which includes principal investigator).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Food Ketogenic Diet (WFKD) (Experimental): Following a 3 week whole food diet run-in, participants will reduce their carbohydrate intake to 30-50g per day to achieve nutritional ketosis.
  Interventions: Behavioral: Whole Food Ketogenic Diet
- Whole Food Diet (WFD) (Active Comparator): Participants will consume a whole-food diet focused on improving diet quality based on the NOVA classifications of unprocessed or minimally processed foods/ingredients (removal of NOVA category 4 foods from diet). This diet is high carbohydrate (45-65% of total energy coming from carbohydrate).
  Interventions: Behavioral: Whole Food Diet

INTERVENTIONS:
Behavioral: Whole Food Ketogenic Diet — Education around immediate changes to improve diet quality and barriers to dietary behaviour change. Participants will consume a whole-food diet focused on improving diet quality based on the NOVA classifications of unprocessed or minimally processed foods/ingredients (removal of NOVA category 4 foods from diet). This group will focus on the consumption of low-energy, nutrient dense whole foods with a targeted carbohydrate intake of 30-50g per day to achieve nutritional ketosis. The WFKD will adjust carbohydrate level for the individual participant to achieve average blood/urinary ketone levels of between 0.5 and 3.0 mmol/L (tested for objective feedback using a mix of urinary ketone sticks and finger prick blood measures).
  Other Names: WFKD; Keto Diet; ketogenic diet
  Arms: Whole Food Ketogenic Diet (WFKD)
Behavioral: Whole Food Diet — Education around immediate changes to improve diet quality and barriers to dietary behaviour change. Participants will consume a whole-food diet focused on improving diet quality based on the NOVA classifications of unprocessed or minimally processed foods/ingredients (removal of NOVA category 4 foods from diet). This diet is high carbohydrate (45-65% of total energy coming from carbohydrate, 20-35% from fat and 15-25% from protein) based on the Australian dietary guidelines focusing on the consumption of low-energy, nutrient dense whole foods. The higher carbohydrate diet reflects current contemporary 'standard care' dietary recommendations as outlined by the National Health and Medical Research Council's Australian Dietary Guidelines, and therefore represents the most appropriate control diet to compare to the effects of the proposed intervention.
  Other Names: WFD; Minimally Processed Diet
  Arms: Whole Food Diet (WFD)

SUMMARY:
The aim of this project is to learn about how a change in diet will affect sleepiness, quality of life and metabolic health in people living with narcolepsy and idiopathic hypersomnia. The dietary changes we will be testing are well researched and safe in a wide range of patient groups (such as in obesity, type one and two diabetes, cancer and dysfunction related to the nervous system) but has not been researched in conditions of hypersomnolence such as narcolepsy and idiopathic hypersomnia. It is important to test adjunct therapies and lifestyle changes such as dietary interventions to ensure that people living with hypersomnolence have a range of options in addition to medications, to improve their health.

If effective, this project will be tested in more people and may become a part of routine patient care. These dietary approaches have been shown to improve health and quality of life in people living with chronic pain, neurological conditions such as epilepsy and have been shown to be safe in these populations as well as people living with type one diabetes. This is a new area of research for people living with hypersomnolence.

DETAILED DESCRIPTION:
The primary objectives of COMPANION are:

• To determine the feasibility and tolerability of a 12-week whole-food ketogenic diet (WFKD) compared to an isocaloric standard whole-food diet (WFD) in participants with hypersomnolence (HS) as defined by the RE-AIM Framework.

The secondary objectives are:

* To determine whether a WFKD achieves greater improvements in disease relevant sleep outcomes including excessive daytime sleepiness, reduced duration of sleep onset latency and psychomotor vigilance compared to an isocaloric WFD in participants with HS.
* To determine whether a WFKD achieves greater improvements in objective metabolic health outcomes and subjective quality of life outcomes compared to an isocaloric WFD in participants with HS.
* To determine whether patients prefer a combination of dietary intervention and medication or unique dietary intervention compared to traditional medication only treatments in their lived experience.
* To better understand the context for implementation of both dietary interventions, determining the barriers and facilitators to widespread implementation of the dietary intervention.

A prospective, mixed methods, randomised, single-centre, controlled trial (Hybrid Type 1) with two parallel groups comparing the feasibility of a WFKD to a WFD stratified by patient diagnosis of NT1, NT2 or IH. This project will determine whether patients with persistent HS can feasibly sustain dietary changes in addition to usual care, and if so, whether improvements in symptoms of daytime sleepiness, metabolic health and quality of life outcomes can be enhanced with a WFKD. At the core of this project is the delivery of a 12-week dietary intervention, in which all patients will be initially allocated to a WFD for three weeks. At the commencement of week four, participants will be randomised to either maintain consumption of this WFD or combine with carbohydrate restriction to form a WFKD for the remaining nine weeks.

The inclusion of a three-week run-in period for all patients provides confidence to the design that patients entering randomisation can engage with dietary change, and thus will provide our first indicator of feasibility. The WFD group from this point on will serve as a comparator in this randomised clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Evidence (from multiple sleep latency test, 24-hour polysomnography, or actigraphy) of diagnosis of narcolepsy type 1, narcolepsy type 2 or idiopathic hypersomnia that meets ICSD-3 criteria.
* For the NT1 subtype, patients must have been screened positive for the HLA DQB10602 genotype.
* Body mass index >18.5 kg/m2
* 18 years or over
* Be willing to be involved in dietary change that may include animal protein and fat.
* Be willing to monitor ketones via finger-prick and urinary dipstick.
* Habitual diet is a standard diet consuming a moderate or high carbohydrate level (defined for the study as above 130g carbohydrate/day).
* Willingness to provide informed consent and willingness to participate and comply with the study requirements.
* Access to a computer, laptop, tablet, or smartphone and stable internet access.
* Proficient comprehension of English language (able to independently read information sheet) and availability of a support person during consultations if English comprehension is challenged.

Exclusion Criteria:

* Body mass index <18.5 kg/m2, history of an eating disorder with an EDE-Q score greater than 3.
* Participants who have sustained significant weight loss in the last 3 months (>5% change in total body weight).
* Previous bariatric surgery or current prescription of weight loss medication.
* Diagnosis of unstable psychiatric disorders (excluding anxiety or depression).
* Cognitive impairment that limits ability to understand the study requirements or provide informed consent.
* Physical impairment that limits ability to meet the study requirements.
* Non-English speaking and inability to read the Participant Information Sheet.
* No access to stable internet and device on which to participate in telehealth consultations and complete study questionnaires.
* Person lactating, pregnant or of childbearing potential who are not willing to avoid becoming pregnant during the study period.
* Habitual diet is currently low carbohydrate/ketogenic (defined for the study as <130g carbohydrate/day based on screening 24 food hour recall).
* Habitual diet excludes animal products (e.g. Vegan diet).
* Laboratory parameters that may indicate alternate catalyst for hypersomnolence in the opinion of the study physician, including abnormal: full blood count, thyroid function, Epstein-Barr Virus, erythrocyte sedimentation rate, cortisol, antinuclear antibodies, extractable nuclear antigen test, positive rheumatoid factor, Antistreptolysin O positive, Iron studies or multiple biochemistry panel.
* Participants who have changed their medication prescription or dose within the preceding 4 weeks.
* Participants with inherited metabolic disorders, prior history of hypoglycaemia or insulinoma
* Participants with insulin dependent Type 1 or Type 2 diabetics prescribed insulin which may interfere with the participant's ability to meet the study requirements.
* Participants with uncontrolled medical conditions or patients with significant medical co-morbidities who in the opinion of the study physician, would be at risk of adverse health consequences due to the study intervention (e.g. poorly controlled type 2 diabetic patients who are not prescribed insulin)
* Current cancer diagnosis (excluding skin cancers or benign cancers)
* Current active enrolment in a pharmaceutical or intervention based clinical trial or participant who may have received an investigational new drug within the last 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility - using quantitative measures of feasibility | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  A suite of quantitative measures of feasibility (i.e. recruitment rate related to the number of patients considered for eligibility, screened, enrolled and the time frames associated with reaching the target sample size) will be measured during the 3-month dietary intervention. The primary outcomes will be triangulated with qualitative interviews to provide an overall assessment of trial feasibility. Results at 12 weeks and baseline will be compared.
Feasibility - using quantitative measures of tolerability | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  A suite of quantitative measures of tolerability (measured by dietary protocol adherence, rate of attrition during both the run in and intervention phase and quantity and nature of adverse events) will be measured during the 3-month dietary intervention. The primary outcomes will be triangulated with qualitative interviews to provide an overall assessment of trial feasibility. Results at 12 weeks and baseline will be compared.
Feasibility - using quantitative measures of compliance | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  A suite of quantitative measures of compliance (measured by capillary and urinary ketones and food diaries) will be measured during the 3-month dietary intervention. The primary outcomes will be triangulated with qualitative interviews to provide an overall assessment of trial feasibility. Results at 12 weeks and baseline will be compared.

SECONDARY OUTCOMES:
Sleep Outcomes - average sleep onset latency | From baseline visit in week 0 to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  The key sleep efficacy outcome is the average sleep onset latency in minutes measured across 5 trials of the maintenance of wakefulness test (MWT) at 12 weeks compared with baseline.
Sleep Outcomes - markers of sleep micro-architecture | From baseline visit in week 0 to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Markers of sleep micro-architecture during PSG including sleep onset latency, REM onset latency, sleep duration, sleep efficiency measured at 12 weeks compared with baseline.
Sleep Outcomes - Narcolepsy Severity Scale (for NT1 and NT2) | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Change in Narcolepsy Severity Scale measured at 12 weeks compared with baseline and 3 weeks.
  The Narcolepsy Severity Scale is a 15-item self-reported outcome measure validated for use in NT1 patients. It evaluates the severity, frequency, and impact of the 5 main narcolepsy symptoms (EDS, cataplexy, hallucinations, sleep paralysis, and disrupted night-time sleep). Total score ranges from 0 to 57, with higher scores indicating more severe symptoms. Except for cataplexy, these narcolepsy symptoms are also relevant for some NT2 patients, and thus, we will use the Narcolepsy Severity Scale in both NT1 and NT2 patients.
Sleep Outcomes - Idiopathic Hypersomnia Severity Scale (for IH) | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Change in Idiopathic Hypersomnia Severity Scale measured at 12 weeks compared with baseline and 3 weeks.
  The Idiopathic Hypersomnia Severity Scale is a self-reported measure validated in patients with IH. It is a 14-item questionnaire that measures aspects of night-time and daytime sleep symptoms and the sleep inertia related to each, as well as impaired daytime functioning due to hypersomnolence. Symptom frequency, intensity, and consequences are rated using a 3- or 4-point scale. Total score ranges from 0 to 50, with higher scores indicating more severe and frequent symptoms.
Sleep Outcomes - weekly cataplexy rate | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Weekly cataplexy rate (in patients with NT1 only): patients will be asked the number of cataplectic events each day (and description if full or partial events) alongside the sleep diary in week 12 (prior to the final visit), compared to the week prior to baseline, and during week 3 (the week prior to randomisation).
Sleep Outcomes - Karolinska Sleepiness Scale | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Karolinska Sleepiness Scale (KSS): Participants will be asked to rate their sleepiness before each MWT trial using the KSS, a 9-point Likert scale designed to assess their state of sleepiness at any given time measured at 12 weeks compared to baseline. A higher KSS score indicates a higher level of subjective sleepiness.
Sleep Outcomes - Epworth Sleepiness Scale | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Change in Epworth Sleepiness Scale: Participants will be asked to rate on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities to provide an indication of their daytime sleepiness measured at 12 weeks compared to baseline and 3 weeks. Higher scores suggest higher levels of excessive daytime sleepiness.
Sleep Outcomes - Psychomotor Vigilance Task (PVT) | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  The PVT will be used to assess sustained attention via a simple reaction time task. The device is a hand-held box with a red-light emitting diode display of a three-digit millisecond counter (PVT-192, Ambulatory Monitoring Inc, Ardsley, NY, USA). Participants are instructed to respond as fast as possible when they first see a visual stimulus appear. The time taken to respond to the stimulus is displayed in milliseconds (ms). During each 10-minute PVT session, visual stimuli appear at variable intervals between 2 to 10 seconds. The PVT response variables to be analysed are: a) mean reciprocal reaction time (RT); b) mean of the fastest 10% of RTs; c) mean reciprocal of slowest 10% of RTs; and, d) number of lapses (response time >500ms). Tests will take place after each MWT trial.
Exploratory Sleep Outcomes - quantitative analysis of the EEG from PSG data | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Quantitative analysis of the EEG from PSG data for assessment of sleep microarchitecture including power spectral analysis across all frequencies throughout the entire sleep period and separately in REM and non-REM sleep, K-complexes, and sleep spindles. These will be measured at 12 weeks compared to baseline.
Cardio-metabolic and Quality of Life Outcomes - high sensitivity C-reactive protein (hs-CRP) | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  The key metabolic efficacy outcome is the blood pathology-based measure of high sensitivity C-reactive protein (hs-CRP) at 12 weeks compared with baseline.
Cardio-metabolic and Quality of Life Outcomes - 36-Item Short Form Survey summary scores | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  The key quality of life efficacy outcome is the 36-Item Short Form Survey (SF-36) summary scores (Physical Component Summary score and the Mental Component Summary) at 12 weeks compared with baseline.
  The SF-36 is a 36-item, patient-reported measure of health status consisting of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Cardio-metabolic and Quality of Life Outcomes - laboratory blood analyses | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Laboratory Analyses for metabolic risk, inflammatory markers and hormones: A 25mL fasted blood sample will be collected by a trained professional at a commercial laboratory at baseline and at 3 months to assess cardio-metabolic risk and inflammatory status at baseline, end of week 3 and week 12. Outcome measures will include hs-CRP, erythrocyte sedimentation rate (ESR), fasting glucose and insulin [HOMA-IR for insulin resistance], blood lipids and lipoproteins and liver function.
Cardio-metabolic & Quality of Life Outcomes - anthropometry and vitals data | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Anthropometry and vitals data: weight, waist circumference, neck circumference, heart rate and blood pressure will be measured at baseline and 12 weeks.
Cardio-metabolic & Quality of Life Outcomes - assessment of mood and quality of life using 36-Item Short Form Survey | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Assessment of mood and quality of life will be assessed at baseline, 3 weeks and 12 weeks using the SF-36: The 36-Item Short Form Survey (SF-36) is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status consisting of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Cardio-metabolic & Quality of Life Outcomes - assessment of mood and quality of life using Hospital Anxiety and Depression Scale | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Assessment of mood and quality of life will be assessed at baseline, 3 weeks and 12 weeks using the Hospital Anxiety and Depression Scale (HADS): The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher scores indicate higher levels of anxiety or depression.
Cardio-metabolic & Quality of Life Outcomes - assessment of mood and quality of life using EQ-5D-5L | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Assessment of mood and quality of life will be assessed at baseline, 3 weeks and 12 weeks using the EQ-5D-5L: The EQ-5D questionnaire comprises two parts. The first is the EQ-5D descriptive system, respondents are asked to tick boxes to indicate the level of problem respondents experience on each of the five dimensions. The combination of these ticks under each dimension describes that person's EQ-5D self-reported health state. The second part of the questionnaire is the EQ VAS, so called because it incorporates a Visual Analogue Scale. This captures the respondent's overall assessment of their health on a scale from 0 (worst health imaginable) to 100 (best health imaginable).
Cardio-metabolic & Quality of Life Outcomes - assessment of mood and quality of life using Clinical Global Impression | At the end of 12 weeks for the last enrolled participant.
  Assessment of mood and quality of life will be assessed at 12 weeks only using the Clinical Global Impression Instrument: rating scales are measures of symptom severity, treatment response and the efficacy of treatments. It is a brief 3-item observer-rated scale undertaken by the clinician at the end of an intervention period. It consists of a severity scale, an improvement scale and an efficacy index. Severity of illness is rated on a 7-point scale, ranging from 1 (normal) through to 7 (amongst the most severely ill patients). Global improvement is rated on a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse). Efficacy index describes both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side-effects) to 16 (unchanged or worse and side-effects outweigh the therapeutic effects).
  Each component of the CGI is rated separately; the instrument does not yield a global score.
Demographics & diagnostic history | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  The following information will be collected via a survey at the time of enrolment: age, sex, health status, evidence of diagnosis as per inclusion criteria, time since diagnosis and medications relating to participant HS condition.
  The following demographics will be measured at the baseline and 12 week visits: height (baseline only), weight, waist circumference, office blood pressure.
Adherence and lived experience during intervention - diet satisfaction | From the end of 3 weeks to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through surveys including diet satisfaction: convenience, flexibility and enjoyment. The 45-item Dietary Satisfaction Questionnaire (DSat-45) uses seven scales to assess characteristics that influence diet satisfaction: Healthy Lifestyle, Convenience, Cost, Family Dynamics, Preoccupation with Food, Negative Aspects, and Planning and Preparation. The items are assessed using five responses ranging from 'Disagree Strongly' to 'Agree Strongly', which are scored from 1 to 5. Items are reverse-scored if necessary, so that higher scores indicate greater diet satisfaction, and scale scores are created by averaging scores across items. A Total Diet Satisfaction score is also calculated by averaging all item scores. This will be measured at the end of 3 and 12 weeks only.
Adherence and lived experience during intervention - macronutrient/micronutrient change | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through diaries including macronutrient/micronutrient change: Measurement of increased nutrient density or changes in macronutrient distribution assessed using 24-hour food recalls. Participants will use the ASA24 (2016, Australian version) developed by the National Cancer Institute (USA) and adapted to the Australian context by Australian researchers. It is a self-administered 24-hour dietary recall tool that enables a multiple, automatically coded food diary. It provides food choices based on the Australian Food, Supplement and Nutrient database (AUSNUT) 2011-13. Data will be collected prior to each telehealth consultation. This will be measured at baseline 3, 4, 6, 8, 10 and 12 weeks only.
Adherence and lived experience during intervention - dietary adherence measured by blood ketosis level | From the baseline visit in week 0 to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through objective measures of compliance including dietary adherence measured by ketosis level: The level of ketones achieved and duration of ketone levels within the nutritional ketosis range (0.5-3mmol/L) as ascertained by a finger-prick test using an Abbott Freestyle Optium Neo (https://www.youtube.com/watch?v=X819_lhKpw0) and urinary dipsticks. All participants will measure morning and evening capillary ketones two days per week.
Adherence and lived experience during intervention - dietary adherence measured by urine ketosis level | From the baseline visit in week 0 to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through objective measures of compliance including dietary adherence measured by ketosis level: The level of ketones achieved and duration of ketone levels within the nutritional ketosis range (0.5-3mmol/L) as ascertained by urinary dipsticks. All participants will measure afternoon/evening urinary ketone levels four times per week.
Adherence and lived experience during intervention - habitual actigraphy sleep-wake data | From week -1 to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through objective measures of compliance including habitual sleep-wake data: will be collected to describe temporal patterns of sleep and activity. This will be measured using 7-day actigraphy monitors (GeneActiv wrist watch) in the week prior to baseline visit, the end of week 3 and during week 12.
Adherence and lived experience during intervention - habitual sleep diary sleep-wake data | From week -1 to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through diaries including habitual sleep-wake data: will be collected to describe temporal patterns of sleep and activity. This will be measured using a modified Karolinska sleep diary in the week prior to baseline visit, the end of week 3 and during week 12.
Adherence and lived experience during intervention - Patient Reported Experience Measures - Longitudinal PREM | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through surveys including Patient Reported Experience Measures: collect information about the experience of health services, and the outcomes of health services, as described by patients. At baseline, the Longitudinal PREM will be collected. This survey collects information related to adults receiving care that extends over a long period of time and is seen as a longitudinal capture of a person's experience.
Adherence and lived experience during intervention - Patient Reported Experience Measures - Patient Assessment of Chronic Illness Care | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through surveys including Patient Reported Experience Measures: collect information about the experience of health services, and the outcomes of health services, as described by patients. At baseline, the Patient Assessment of Chronic Illness Care (PACIC) will be collected. This survey collects information related to adults receiving care that extends over a long period of time and is seen as a longitudinal capture of a person's experience.
Adherence and lived experience during intervention - Patient Reported Experience Measures - Outpatient PREM | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Aim to characterise participant behaviour and lived experience through surveys including Patient Reported Experience Measures: collect information about the experience of health services, and the outcomes of health services, as described by patients. At 12 weeks, the Outpatient PREM question set will be collected. This survey collects data capturing the patients' experiences of outpatient clinics and services.
Qualitative Data - semi-structured interviews | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Qualitative data will be collected through semi-structured interviews related to the patient experience.
  Thematic analysis of these qualitative interviews will be conducted at three key timepoints during the intervention. These will align with:
  * The commencement of intervention (to characterise the patient lived experiences and expectations),
  * The end of the three-week whole food run in period (dietary change evaluation),
  * The end of the twelve-week intervention (process evaluation).
Qualitative Data - overall project evaluation | From enrolment to the completion of the last study visit at the end of 12 weeks for the last enrolled participant.
  Overall project evaluation will be assessed using the implementation plan using the RE-AIM Framework and the CFIR framework.
  The implementation plan will evaluate the randomized controlled trial in synchrony with thematic analysis of a series of qualitative interviews conducted at three key timepoints during the intervention. These will align with the commencement of intervention (to characterise the patient lived experiences and expectations), at the end of the three-week whole food run in period (dietary change evaluation), and at the end of the twelve-week intervention (process evaluation). These interviews will provide a platform to better understand the patient experience during the intervention and will guide future iterations of the program.
  The evaluation methodology will use a combination of the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) and CFIR (Consolidated Framework for Implementation Research) dissemination and implementation frameworks.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Machan, PhD, Principal Investigator — University of Sydney; Sheila Sivam, PhD; MD; FracP; BSc (Med), Principal Investigator — Royal Prince Alfred Hospital and University of Sydney
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No